CLINICAL TRIAL: NCT06612788
Title: A Feasibility Clinical Trial of Exablate for Low Intensity Focused Ultrasound Neuromodulation in Patients With Opioid Use Disorder (OUD) and/or Other Substance Abuse Disorders (SUDs)
Brief Title: Exablate for LIFU Neuromodulation in Patients With Opioid Use Disorder (OUD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUD001; UH3DA047714-04S1 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-09

CONDITIONS: Opioid Use Disorder
Keywords: Narcotic-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Opioid-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sham/Active ExAblate Treatment Stage 1 and 2 (Other): Subject will undergo both Treatment 1 (sham) and Treatment 2 (with enhanced intensity). Subjects are blinded to the order of the sham vs active treatment.
  Interventions: Device: Exablate Model 4000 Type 2.0/2.1

INTERVENTIONS:
Device: Exablate Model 4000 Type 2.0/2.1 — There are two treatment stages. In both stages, the subject will receive both the sham and active ExAblate treatment, and be evaluated for 90 days post-treatment for adverse events. During Stage 1 the subject will receive the moderate intensity Exablate LIFU procedure. During Stage2, the subject will receive the enhanced intensity ExAblate LIFU procedure. The subjects are blinded as to the order of the sham vs active treatment.

SUMMARY:
The purpose of this clinical trial is to investigate Low Intensity Focused Ultrasound (LIFU) using the Exablate® Model 4000 Type 2.0/2.1 as an adjunctive neuromodulatory treatment for OUD (Opioid Use Disorder) by assessing its safety and tolerability in subjects with OUD.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females, age 18 - 60 years old
* Subject meets DSM-5 criteria for OUD and/or other SUDs including alcohol (assessed via the SCID-5) of at least two years duration
* Subject is currently receiving outpatient treatment from the WVU Comprehensive Opioid Addiction Treatment Program (COAT), Intensive Outpatient Program (IOP) or any other program which implements the COAT model; residential or inpatient treatment from the WVU Center for Hope and Healing or an affiliated WVU hospital; or receiving outpatient/inpatient/residential treatment from similar programs that are well known to the research team. If the subject is prescribed medication for AUD or OUD (e.g. buprenorphine-naloxone, naltrexone), they will be on a stable dose of the medication for the 7 days prior to the procedure. Stable is defined as within the therapeutic range but does not require same exact dose for 7 days.
* Subject has been off opioids and other illicit substances, except for cannabis, confirmed via urine toxicology screen
* The NAc is apparent on MRI such that treatment targeting can be performed directly (visible on MRI) and indirectly (using other anatomical structures for measurements)
* Subject is able to communicate sensations during the Exablate Transcranial procedure
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all study visits
* Subject is able to make own medical decisions as determined by the clinical team
* Subject has signed and received a copy of the approved informed consent form

Exclusion Criteria:

* Subjects who are taking medications which may adversely interact with MOUD (See Appendix B for full list). Being on one of these medications would not automatically exclude a participant from study participation, does not automatically exclude a prospective subject from study participation. If a prospective or current subject is taking any medication listed in Appendix B, the study investigator is responsible for determining whether the subject is eligible for inclusion or continued study participation.
* Subject with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices
* Subject with known intolerance or allergies to the MRI contrast agent gadolinium (GADOVIST®)
* Subject who are unable or unwilling to tolerate the required prolonged stationary position during treatment (approximately 2-3 hours)
* More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
* Subject with implanted objects in the skull or the brain
* Subject diagnosed with advanced kidney disease or on dialysis
* Subject with impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
* Subject with known unstable cardiac status or severe hypertension including:

Documented myocardial infarction within six months of enrollment Unstable angina on medication Unstable or worsening congestive heart failure Left ventricular ejection fraction below the lower limit of normal History of a hemodynamically unstable cardiac arrhythmia Cardiac pacemaker Severe hypertension (diastolic BP > 100 on medication)

* Subject with history of abnormal bleeding, hemorrhage, or coagulopathy
* Subject receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Abnormal coagulation profile (PLT < 100,000/μl), PT (>13.9 sec) or PTT (>37.5 sec), and INR > 1.2. If values are outside the range of normal limits, any clinically significant value may be excluded as determined by a study investigator.
* Subject with cerebrovascular disease as determined by MRI according to the Fazekas criteria. Grades II and III on the Fazekas scale should be excluded
* Past or present diagnosis of schizophrenia, psychotic disorder, bipolar disorder, or untreated depression other than one determined to be substance induced (assessed via SCID-5)
* Score of greater than 17 on the Hamilton Depression Rating Scale (HAM-D) or increased risk of suicide based on any positive response regarding passive or active suicidal ideation with or without intent over the past 3 months or lifetime history of active suicidal ideation with intent on the Columbia-Suicide Severity Rating Scale (C-SSRS) at baseline
* History of suicide attempt
* Parental history of completed suicide
* Subject meet the criteria for Cluster A or B Personality Disorders (assessed via SCID-5-PD)
* Diagnosis of dementia or any other disorder which has led to a clinically significant cognitive impairment (assessed via NIHTB-CB)
* Subject with brain tumors
* Subject with chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area
* Any known CNS infection or infection with the Human Immunodeficiency Virus (HIV) or Hepatitis C (HCV). A diagnosis of Hepatitis C (HCV) alone is not exclusionary as long as hepatic function laboratory values are deemed not clinically significant by a study investigator and are ≤ 1.5 times the upper limit of normal.
* Subject who has had deep brain stimulation or a prior stereotactic ablation of the NAc, basal ganglia or thalamus
* Subject who has been administered botulinum toxins into the arm, neck, or face for 5 months prior to baseline
* Subject who is currently participating in another clinical investigation with an active treatment arm
* Subject unwilling to abstain from illicit substance use during the course of the study
* Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator
* Subject is non-English speaking
* Subject is pregnant or planning to be pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | Post-ExAblate Procedure (Day 0) through 4 Month Follow-Up
  Safety will be assessed by recording all adverse events that are treatment related. Each Adverse Event will be documented for patterns of occurence.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — WVU Rockefeller Neuroscience Institute
Locations (1):
- West Virginia University: Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States